CLINICAL TRIAL: NCT06998342
Title: MOHs Surgery and Adjuvant Short-course Hypofractionated Radiation Therapy With Structured Surveillance for Cutaneous Head & Neck Squamous Cell Carcinoma: a Phase II Pilot Study (MOHSAHRTSS-Study)
Brief Title: MOHs Surgery and Short-Course Radiation Therapy With Structured Follow-Up for Head & Neck Squamous Cell Skin Cancer
Acronym: MOHSAHRTSS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Anker, Radiation Oncologist. Professor, Radiation-Oncology, University of Vermont Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVMCC2410/STUDY00003513
Record Dates: First submitted 2025-05-07; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous Squamous Cell Carcinoma (CSCC)
Keywords: Cutaneous Squamous Cell Carcinoma; Head and Neck Cancer; Neoadjuvant Therapy; Immunotherapy; Surgical Oncology; Clinical Trial; Radiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Risk Cohort (Experimental): Patients meeting moderate-risk criteria will not receive adjuvant radiation therapy but will instead be monitored through regular clinical exams and imaging. This arm evaluates whether active surveillance is a safe alternative to radiation in this population by tracking recurrence rates and overall survival.
  Interventions: Other: Active Surveillance
- High-Risk Cohort (Experimental): Patients classified as high risk will undergo SCRT, consisting of five fractions of radiation therapy over a two-week period. This approach aims to provide effective local control while minimizing treatment burden compared to conventional long-course radiation therapy (typically 30+ fractions over six weeks). The study will assess the efficacy, safety, and long-term outcomes of SCRT, including recurrence rates, toxicity profiles, and patient-reported quality of life.
  Interventions: Radiation: Short course radiation; Other: Active Surveillance

INTERVENTIONS:
Radiation: Short course radiation — The radiation arm in this study involves Short Course Radiation Therapy (SCRT), which consists of 5 fractions delivered twice a week (either Monday/Thursday or Tuesday/Friday).
  Arms: High-Risk Cohort
Other: Active Surveillance — The Active Surveillance arm (Group M) aims to monitor participants with moderate-risk cutaneous squamous cell carcinoma (cSCC) after surgical resection, without immediate intervention unless disease progression occurs. Participants will undergo regular clinical evaluations, physical exams, and skin checks to detect new lesions or signs of recurrence. Imaging, including ultrasound and CT/MRI scans, will be performed every 6 months for up to 3 years to monitor for metastasis or progression. Blood samples will be collected for future biomarker analysis to identify indicators of disease recurrence. Participants will also complete quality of life assessments using the EORTC QLQ-C30 and Skin Cancer Index (SCI) to evaluate the impact of surveillance on their daily lives. If disease progression is detected, radiation therapy may be initiated. The study will track overall survival without initiating radiation, as well as disease progression and quality of life outcomes, to determine if active s

SUMMARY:
The goal of this clinical trial is to evaluate if short-course radiation therapy (SCRT) can effectively treat high-risk cutaneous squamous cell carcinoma (cSCC) and if active surveillance is a safe alternative to radiation for moderate-risk cSCC in adults with head and neck cSCC who have undergone surgery.

The main questions it aims to answer are:

Does short-course radiation therapy (5 treatments over 2 weeks) effectively prevent cancer recurrence in high-risk patients? Can moderate-risk patients be safely monitored with active surveillance instead of receiving radiation?

Researchers will compare:

Short-course radiation therapy (SCRT) for high-risk patients to historical data on long-course radiation to determine effectiveness.

Active surveillance for moderate-risk patients to expected recurrence rates to assess safety.

Participants will:

High-Risk Group (SCRT): Receive short-course radiation therapy and attend follow-up visits.

Moderate-Risk Group (Active Surveillance): Have regular check-ups, including clinical exams and imaging, to monitor for cancer recurrence.

Optionally provide blood samples for future biomarker research.

DETAILED DESCRIPTION:
This clinical trial investigates two approaches for managing cutaneous squamous cell carcinoma (cSCC) of the head and neck following surgical resection, based on patient risk stratification. The study evaluates short-course radiation therapy (SCRT) as a treatment for high-risk cSCC and active surveillance as a potential alternative to radiation therapy for moderate-risk cSCC.

High-Risk Cohort (Short-Course Radiation Therapy - SCRT) Patients classified as high risk will undergo SCRT, consisting of five fractions of radiation therapy over a two-week period. This approach aims to provide effective local control while minimizing treatment burden compared to conventional long-course radiation therapy (typically 30+ fractions over six weeks). The study will assess the efficacy, safety, and long-term outcomes of SCRT, including recurrence rates, toxicity profiles, and patient-reported quality of life.

Moderate-Risk Cohort (Active Surveillance) Patients meeting moderate-risk criteria will not receive adjuvant radiation therapy but will instead be monitored through regular clinical exams and imaging. This arm evaluates whether active surveillance is a safe alternative to radiation in this population by tracking recurrence rates and overall survival.

Study Design and Assessments Participants will be followed for oncologic outcomes (local, regional, and distant recurrence rates), adverse events, functional outcomes, and patient-reported quality of life. Optional blood sample collection will allow for biomarker analysis and potential future translational research.

By stratifying patients based on risk, this trial aims to refine post-surgical management of head and neck cSCC, potentially reducing unnecessary radiation exposure in moderate-risk patients while ensuring effective treatment for high-risk individuals.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed cutaneous squamous cell carcinoma of the head & neck region, defined as extending from vertex of head to supraclavicular region.
* Mohs micrographic surgery with or without further surgery following Mohs to achieve negative margins (i.e. R0 margin status) within 70 days prior to registration
* Appropriate stage for study entry (T1-T3 N0 M0; AJCC 8th ed.) based on the following diagnostic workup:

  * Clinical exam within 60 days prior to registration
  * CT head & neck/soft tissue with IV contrast within 60 days prior to registration or MR face and neck with IV contrast. IV contrast may be held if medically contraindicated.
  * Bilateral neck ultrasound within 60 days prior to registration
* Risk Factors fitting either the High-Risk or Moderate-Risk Categories:

  * Risk Factor Definitions

Major Risk Factors: Microscopic Extensive PNI (defined as PNI for >3 nerves with all involved nerves either >0.1 mm in size and/or deeper than the dermis), Gross PNI (defined as perineural spread evidenced on by MRI imaging, with cranial nerve deficit, or both), Size >6 cm, or Recurrent disease status post prior Mohs

Moderate-Risk Factors: Poor differentiation, 4-6 cm, PNI (defined as >0.1 mm in size)

BWH Risk factors: >2 cm, poor differentiation, deep invasion, PNI (>0.1 mm in size)

• BWH: T2a = 1 risk factor; T2b = 2-3 risk factors, T3 = 4 risk factors

High-Risk Group (Group H) Any 1 major OR 2-3 moderate OR BWH T3

Moderate-Risk Group (Group M) BWH T2b not meeting criteria for High-Risk.

Exclusion Criteria:

* Patients receiving any other investigational agents.

Patients pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Serious medical comorbidities that, in the opinion of the radiation oncologist, would prevent participation in this study.

Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for different cancer(s) is allowable

Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields

Actively receiving systemic cytotoxic chemotherapy, immunosuppressive, anti-monocyte or immunomodulatory therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Exploring the Efficacy of Adjuvant Hypofractionated Radiation Therapy in High-Risk cSCC Head and Neck Patients: A Comparison of 2-Year Locoregional Recurrence Rates | 2 years
  To explore the potential efficacy of adjuvant hypofractionated radiation therapy (SCRT) in high-risk cutaneous squamous cell carcinoma (cSCC) head and neck patients by examining the 2-year locoregional recurrence rate (LRR) and comparing it to historical controls who received standard long-course radiation therapy (LCRT). Considering the variability in LRR among patients eligible for SCRT, the researchers aim to investigate whether a 2-year LRR <25% could be achieved.

SECONDARY OUTCOMES:
2-Year Locoregional Recurrence Rate (LRR) in Moderate-Risk SCC Patients | 2 years
  To assess the 2-year rate of locoregional recurrence (LRR) in moderate-risk patients undergoing active surveillance, compared to historical controls. Unit of Measure: Percentage of participants with locoregional recurrence.
2-Year Overall Survival (OS) in High-Risk SCC Patients Receiving SCRT | 2 years
  To evaluate overall survival at 2 years in high-risk patients treated with short-course radiation therapy (SCRT), compared to historical controls who received long-course radiation therapy (LCRT). Unit of Measure: Percentage of participants alive at 2 years.
Health-Related Quality of Life (HRQoL) in High-Risk SCC Patients as Measured by EORTC QLQ-C30 | 3 years
  To assess overall health-related quality of life using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) in patients receiving SCRT or active surveillance. This validated questionnaire includes subscales for physical, emotional, and social functioning, among others. Unit of Measure: Score on scale from 0 to 100; higher scores on functioning scales and global health indicate better outcomes; higher scores on symptom scales indicate worse symptoms.
2-Year Overall Survival (OS) in Moderate-Risk SCC Patients | 2 years
  To assess overall survival (OS) at 2 years in moderate-risk patients undergoing active surveillance. OS is defined as time from surgery to death from any cause. Unit of Measure: Percentage of participants alive at 2 years.
2-Year Disease-Specific Survival (DSS) in Moderate-Risk SCC Patients | 2 years
  To assess disease-specific survival (DSS) at 2 years. DSS is defined as time from surgery to death attributed to cutaneous squamous cell carcinoma (cSCC). Unit of Measure: Percentage of participants who survive without dying from cSCC
Local Recurrence Rate (LR) in Moderate-Risk SCC Patients | 2 years
  To assess the incidence of local tumor recurrence in moderate-risk patients undergoing active surveillance. To assess the incidence of local tumor recurrence in moderate-risk patients undergoing active surveillance.
Regional Recurrence Rate (RR) in Moderate-Risk SCC Patients | 2 years
  To assess the incidence of regional tumor recurrence (e.g., nodal) in moderate-risk patients. Unit of Measure: Percentage of participants with regional recurrence
Distant Metastasis Rate (DMR) in Moderate-Risk SCC Patients | 2 years
  To assess the incidence of distant metastasis at 2 years. Unit of Measure: Percentage of participants with distant metastasis
Total Relapse Rate (TRR) in Moderate-Risk SCC Patients | 2 years
  To assess the 2-year total relapse rate (local, regional, or distant) in moderate-risk patients. Unit of Measure: Percentage of participants with any form of relapse
Rate of Resectability at Recurrence in Moderate-Risk SCC Patients | 2 years
  To assess the proportion of participants with resectable disease upon recurrence. Unit of Measure: Percentage of recurrences deemed resectable
2-Year Disease-Specific Survival (DSS) in High-Risk SCC Patients Receiving SCRT | 2 years
  To evaluate disease-specific survival at 2 years in high-risk patients treated with SCRT, compared to historical controls. DSS is defined as death due to cSCC. Unit of Measure: Percentage of participants surviving without death from cSCC.
Local Recurrence Rate (LR) in High-Risk SCC Patients Receiving SCRT | 2 years
  To evaluate the local recurrence rate at 2 years in high-risk patients treated with SCRT, compared to historical controls treated with LCRT. Unit of Measure: Percentage of participants with local recurrence.
Regional Recurrence Rate (RR) in High-Risk SCC Patients Receiving SCRT | 2 years
  To evaluate the regional recurrence rate at 2 years in high-risk patients treated with SCRT, compared to historical controls treated with LCRT. Unit of Measure: Percentage of participants with regional recurrence.
Distant Metastasis Rate (DMR) in High-Risk SCC Patients Receiving SCRT | 2 years
  To evaluate the distant metastasis rate at 2 years in high-risk patients treated with SCRT, compared to historical controls. Unit of Measure: Percentage of participants with distant metastases
Unit of Measure: Percentage of participants with distant metastases | 2 years
  To evaluate the total relapse rate at 2 years (local, regional, or distant) in high-risk patients treated with SCRT, compared to historical controls treated with LCRT. Unit of Measure: Percentage of participants with any recurrence.
Rate of Resectability at Recurrence in High-Risk SCC Patients Receiving SCRT | 2 years
  To assess the proportion of patients whose recurrence was considered surgically resectable. To assess the proportion of patients whose recurrence was considered surgically resectable.
Skin Cancer-Specific Quality of Life in High-Risk SCC Patients as Measured by the Skin Cancer Index (SCI) | 3 years
  To evaluate quality of life specific to skin cancer using the Skin Cancer Index (SCI), which includes domains such as emotional, social, and appearance-related concerns. Unit of Measure: Score on scale from 0 to 100; higher scores indicate better quality of life.
Patient-Reported Cancer Care Burden as Measured by the Patient Experience Survey (PES) | 3 years
  To assess cancer care-related burdens such as travel, cost, and logistical challenges using the Patient Experience Survey (PES), a custom questionnaire including both Likert-scale and yes/no questions. Unit of Measure: Percentage of patients reporting specific concerns (e.g., % worried about cost, % concerned about transportation).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized patient related data will be incorporated into publications and will be made available to other investigators at reasonable request.